CLINICAL TRIAL: NCT06542185
Title: Investigation of Self-Efficacy Levels of Cardiovascular Surgery Intensive Care Unit Nurses on Safe Blood and Blood Product Transfusion
Brief Title: Self-Efficacy Levels of Nurses on Safe Blood and Blood Product Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Arzu Bahar, Yüksek Ihtisas University, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ABAHAR-003
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: To Evaluate the Effect of Online Education on Nurses' Self-efficacy Regarding Blood Transfusion
Keywords: nurse; blood transfusion; To evaluate the effect of online education on nurses' self-efficacy regarding blood transfusion practices.

STUDY DESIGN:
Intervention Model Description: Parallel Assignment a clinical trial with experimental and control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online education (Experimental): - Nurses' self-efficacy levels regarding safe blood transfusion practices will be measured with the Safe Blood and Blood Products Transfusion Self-Efficacy Scale (SBT-SES). SBT-SES pre-tests will be applied to the control and intervention groups, and online training on safe blood transfusion prepared by the researcher will be provided to the intervention group. After the training given to the intervention group, SBT-SES post-tests will be applied to both the intervention and control groups.
  Interventions: Other: online education
- control (No Intervention): No training will be given, only the Blood Products Transfusion Self-Efficacy Scale (SBT-SES) pre-test and post-test will be conducted.

INTERVENTIONS:
Other: online education — online education
  Arms: online education

SUMMARY:
A quasi-experimental study was conducted in a pre-test-post-test design to investigate the self-efficacy levels of nurses working in a cardiovascular surgery Intensive Care Unit regarding safe blood and blood product transfusion and the effects of online training.

DETAILED DESCRIPTION:
Blood transfusion is a life-saving and therapeutic procedure, but it also carries high risks. Nurses have the greatest responsibility in preventing complications related to blood transfusion. To maintain safe practice standards, healthcare institutions need to use national transfusion guidelines and establish blood banks/transfusion laboratories, transfusion protocols, and hemovigilance teams. From the moment the blood is collected from the donor to the end of the transfusion, administering the right blood to the right patient, storing the blood appropriately, monitoring the patient for signs of reactions during the procedure, and having sufficient knowledge and skills on precautions to be taken when complications develop are the responsibilities of nurses regarding transfusion. For nurses to fulfill their duties in this regard, they must have up-to-date knowledge, skills, and competence. Since CVS intensive care clinics are where blood transfusion is performed most frequently, it is of particular importance that the nurses working in these units have sufficient knowledge on the subject and are strengthened in this regard. Based on this situation, the research is planned to determine the self-sufficiency levels of nurses working in the CVS intensive care unit regarding blood transfusion and to contribute to the field by eliminating deficiencies in this regard through training.

ELIGIBILITY:
Inclusion Criteria:

* volunteer nurses

Exclusion Criteria:

* Nurses who did not want to participate in the study

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 20 minutes
  This form, prepared by researchers, includes a total of 13 questions that include nurses' personal and professional characteristics as well as their experiences with blood transfusion (age, gender, professional experience, education, having performed a transfusion, etc.).

SECONDARY OUTCOMES:
Blood Products Transfusion Self-Efficacy Scale (SBT-SES) | 50 minutes
  Blood and Blood Products Transfusion Self-Efficacy Scale contains 49 items. The 5-point Likert type scal. Behavioral Sub-Factor with 16 items; Cognitive Sub-Factor with 14 items; The Attitudinal Sub-Factor consists of 13 items; The Negative Sub-Factor consists of six items. The six items in the negative sub-dimension are reverse and should be reverse-coded during analysis. The minimum score that can be obtained from the total scale is 49 and the maximum score is 245. As the scores obtained from the entire scale and its sub-dimensions increase, it is evaluated that the self-efficacy of nurses for safe blood and blood product transfusion practices increases.

CONTACTS AND LOCATIONS:
Overall Officials: arzu bahar, Principal Investigator — Yüksek Ihtisas University
Locations (1):
- Yüksek Ihtisas University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No